CLINICAL TRIAL: NCT03110822
Title: A Phase 1 Study of Ruxolitinib, Steroids and Lenalidomide for Relapsed/Refractory Multiple Myeloma (RRMM) Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I-RUX-15-04
Record Dates: First submitted 2017-02-27; First posted 2017-04-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
Keywords: Ruxolitinib; Steroids; Lenalidomide; Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ruxolitinib; Lenalidomide; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; methyl prednisolonate

STUDY DESIGN:
Intervention Model Description: There are 4 study parts: Dose escalation and expansion (Study Part 1), Ruxolitinib/Methylprednisolone Arm (Study Part 2), Expanded Eligibility Criteria (Study Part 3), and High Dose (Study Part 4).
  The first 49 subjects will be enrolled into the Ruxolitinib, Lenalidomide and Methylprednisolone treatment arm (Study Part 1).
  Subjects in Study Part 2 will receive Ruxolitinib and Methylprednisolone until confirmed disease progression. Lenalidomide will be added to the treatment once disease progression is confirmed.
  Subjects in Study Part 3 will receive Ruxolitinib, Lenalidomide and Methylprednisolone treatment.
  Subjects in Study Part 4 will receive high-dose Ruxolitinib and Methylprednisolone treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rux Len and Steroid (Experimental): Ruxolitinib Oral Tablet [Jakafi] at 5mg, 10mg or 15mg BID, Lenalidomide Oral at 5mg or 10mg QD and Methylprednisolone Oral at 40mg QOD. (Dose varies during dose escalation portion of the study)
  Interventions: Drug: Ruxolitinib Oral Tablet [Jakafi]; Drug: Lenalidomide; Drug: Methylprednisolone
- Rux and Steroid until progression, then add Len (Experimental): Subject will receive Ruxolitinib Oral Tablet [Jakafi] at 15mg BID, and Methylprednisolone at 40mg QOD until disease progression. Lenalidomide at 10mg QD will be added to the treatment (Ruxolitinib, Methylprednisolone) once disease progression was confirmed.
  Interventions: Drug: Ruxolitinib Oral Tablet [Jakafi]; Drug: Lenalidomide; Drug: Methylprednisolone
- Expanded Eligibility Criteria (Experimental): Subject will receive Ruxolitinib Oral Tablet [Jakafi] at 15mg BID, Lenalidomide at 10mg QD, and Methylprednisolone at 40mg QOD until disease progression.
  Interventions: Drug: Ruxolitinib Oral Tablet [Jakafi]; Drug: Lenalidomide; Drug: Methylprednisolone
- High-dose Ruxolitinib (Experimental): Subject will receive Ruxolitinib Oral Tablet [Jakafi] at 20mg BID and Methylprednisolone at 40mg QOD until disease progression.
  Interventions: Drug: Ruxolitinib Oral Tablet [Jakafi]; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Ruxolitinib Oral Tablet [Jakafi] — Ruxolitinib will be administered on days 1-28 of the treatment cycle.
  Other Names: Ruxolitinib, Jakavi
Drug: Lenalidomide — Lenalidomide will be administered on Days 1-21 of the treatment cycle.
  Other Names: Revlimid
  Arms: Expanded Eligibility Criteria; Rux Len and Steroid; Rux and Steroid until progression, then add Len
Drug: Methylprednisolone — Methyl-prednisolone will be administered on Days 1-28 of the treatment cycle.
  Other Names: Depo-Medrol, Solu-Medrol, Methyl Prednisolonate

SUMMARY:
This is a phase 1, multicenter, open-label study evaluating the safety and efficacy of ruxolitinib, steroids and lenalidomide among MM patients who currently show progressive disease.

DETAILED DESCRIPTION:
Multiple myeloma (MM), a plasma cell dyscrasia, is the most common primary malignancy of the bone marrow.The etiology of myeloma is largely unknown, although genetic predisposition and environmental factors have been speculated. MM arises from malignant plasma cells that clonally expand and accumulate in the bone marrow. These clonal plasma cells produce high levels of monoclonal immunoglobulins. Plasma cell dyscrasias are classified as monoclonal gammopathy of undetermined significance, solitary plasmacytoma, smoldering myeloma, active myeloma, extra-skeletal myeloma, or plasma cell leukemia.

In 2015 an estimated 26,850 adults (14,090 men and 12,760 women) in the United States will be diagnosed with multiple myeloma. It is estimated that 11,240 deaths (6,240 men and 5,000 women) from this disease will occur this year.

In recent years, new and more effective drugs have become available for the treatment of MM. Such drugs have been evaluated together and in combination with older agents, rapidly increasing the number of therapeutic options available to MM patients, and resulting in an improvement in their overall survival (OS) rates. Among the drugs that have been FDA approved specifically for myeloma are the immunomodulatory agents (IMiDs) thalidomide, and its newer analogs lenalidomide and pomalidomide.

IMiDs exert their anti-neoplastic action by affecting various cancer cell functions and the microenvironment, including cytokine production, immune cell function, and in some instances, inflammation, cell proliferation and cell death. The IMiD thalidomide has been found to be effective as an anti-MM agent in one-third of myeloma patients; notably, higher response rates have been observed when combined with steroids. Lenalidomide is an analog of thalidomide that has shown more potent anti-MM activity than thalidomide in preclinical studies, and has been FDA-approved for the treatment of previously untreated as well as relapsed or refractory MM (RRMM) in combination with dexamethasone. Recently, an analog of thalidomide and lenalidomide, pomalidomide, has also been approved for RRMM patients.

The 5-year survival rate for MM patients has increased from 25% in 1975 to 34% in 2003 and is currently closer to 40% due to these newer and more effective treatment options. Unfortunately, even with these newer agents, responses to therapy are transient, and MM remains an incurable disorder with an eventual fatal outcome; and, therefore, new therapies are urgently needed.

JAK2 is an intra-cytoplasmic tyrosine kinase that belongs to the Janus kinase family. JAK kinases play a major role in the transmission of signals from cytokine and growth factor receptors into the nucleus. JAK kinases activate several intracellular signaling proteins, among which the STAT transcription factors are well defined. The JAK/STAT pathway mediates diverse cellular events that affect cell growth, differentiation and cell survival.

Abnormal JAK2 activation has been implicated in several hematological disorders and malignancies. Mutations, gene translocations or cytokines released by bone marrow stromal cells, may all result in aberrant JAK2 activation. The activating JAK2 V617F mutation results in uncontrolled cytokine and growth factor signaling, and is believed to play a key role in the pathophysiology of myeloproliferative neoplasms. Constitutive JAK2 activation through specific chromosomal translocations is thought to contribute to the development of leukemia, lymphoma and multiple myeloma. In MM, elevated levels of cytokines and growth factors such as interleukin-6 (IL 6), vascular endothelial growth factor, insulin-like growth factor-1, basic fibroblast growth factor, IL-1, IL-10, IL-11, IL-15, IL-21, granulocyte macrophage colony stimulation factor, interferon-α, and leukemia inhibitory factor may also contribute to exacerbated JAK2 activation.11 Among these cytokines, IL-6 has been most widely studied and is considered to be a growth and survival factor for myeloma cells. Binding of IL-6 to the IL-6 receptor activates JAK2, which in turn can phosphorylate the IL-6 receptor, thereby augmenting its downstream signaling effects. Thus, pharmacological inhibition of JAK1/2 may be a promising therapeutic strategy for treatment of MM.

In this context, treatment of MM cell lines and patient derived primary MM cells with various JAK1/JAK2, JAK2 and JAK pan specific inhibitors (e.g. INCB16562, CYT387 and TG101209) has been shown to inhibit cell proliferation. Furthermore, JAK inhibitors have demonstrated synergistic activity with established anti MM therapies such as melphalan and bortezomib (CYT387) or melphalan, bortezomib and dexamethasone (INCB16562), in both MM cell lines and patient derived primary MM cells. Sensitization of MM cells to dexamethasone in response to JAK inhibitors may occur through crosstalk between the JAK/STAT pathway and glucocorticoids. In this regard, dexamethasone treatment has been shown to increase STAT3 and the pro survival factor phosphatidylinositol-3 kinase (PI3K) levels in melanoma cells; in turn, PI3K was found to increase STAT3 levels. Prolonged exposure to dexamethasone results in resistance, which could be overcome, at least in part, by JAK/STAT inhibition.

Ruxolitinib is an oral, selective inhibitor of JAK1 and JAK2, and is the only JAK1/2 inhibitor approved by the US FDA for the treatment of intermediate and high-risk myelofibrosis. Pilot experiments carried out in our research laboratory at the Institute for Myeloma and Bone Cancer Research have demonstrated that the JAK2 inhibitor ruxolitinib in combination with lenalidomide and dexamethasone inhibited the proliferation of the MM cell lines U266 and RPMI8226 and primary tumor cells derived from MM patients, and that this inhibition was greater than that achieved with these drugs as single agents. Enhanced anti-tumor activity was also observed when these three drugs were administered together to severe combined immunodeficient mice bearing LAGκ-1A (bortezomib- and melphalan-sensitive) or LAGĸ-2 (bortezomib- and melphalan-resistant) human myeloma tumors, both of which were originally derived from fresh bone marrow biopsies from MM patients. In addition, ruxolitinib as a single agent showed no anti MM effects whereas the combination of this drug with dexamethasone showed enhanced anti-MM effects compared to steroid treatment alone. Finally, an elderly heavily pre treated MM patient with polycythemia rubra vera (PRV), who had previously received single-agent ruxolitinib while progressing from MGUS to MM and then subsequently failed treatment with lenalidomide and methylprednisolone, responded to the addition of low dose ruxolitinib twice daily to these two drugs.

Together, these results suggest that ruxolitinib may overcome lenalidomide and steroid resistance for RRMM patients that are failing therapy from steroids alone or in combination with lenalidomide. Therefore, in this phase 1 trial, the investigators will evaluate the safety and efficacy of ruxolitinib in combination with methylprednisolone and lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible to enroll in this study.

1. Has a diagnosis of MM based on standard criteria as follows:

Major criteria:

1. Plasmacytomas on tissue biopsy.
2. Bone marrow plasmacytosis (greater than 30% plasma cells).
3. Monoclonal immunoglobulin spike on serum electrophoresis IgG greater than 3.5 g/dL or IgA greater than 2.0 g/dL or kappa or lambda light chain excretion greater than 1 g/day on 24 hour urine protein electrophoresis.

Minor criteria:

1. bone marrow plasmacytosis (10% to 30% plasma cells)
2. monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
3. lytic bone lesions
4. normal IgM less than 50 mg/dL, IgA less than 100 mg/dL, or IgG less than 600 mg/dL

Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:

* any 2 of the major criteria
* major criterion 1 plus minor criterion 2, 3, or 4
* major criterion 3 plus minor criterion 1 or 3
* minor criteria 1, 2, and 3, or 1, 2, and 4

  2. Currently has MM with measurable disease, defined as:
* a monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 g/dL and/or
* urine monoclonal protein levels of at least 200mg/24 hours
* for patients without measurable serum and urine M-protein levels, an involved SFLC > 100 mg/L or abnormal SFLC ratio
* for patients with IgD MM, a monoclonal immunoglobulin IgD of at least 1500 mg/L or meet other measurable disease eligibility criteria

  3. Currently has progressive MM

MM patients that are relapsed or have refractory disease from at least 2 regimens or lines of therapy including an IMID and a proteasome inhibitor, are eligible for enrollment provided they fulfill the other eligibility criteria:

* Patients are considered relapsed, when they progress greater than 8 weeks from their last dose of treatment.
* Patients are refractory when they progress while currently receiving the treatment or within 8 weeks of its last dose.

  4. Previous exposure to lenalidomide independent of the response

  5. The patient is not a candidate for a transplant

  6. Understand and voluntarily sign an informed consent form before receiving any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn at any time without prejudice to their future medical care.

  7. Able to adhere to the study visit schedule and other protocol requirements

  8. ECOG performance status of ≤ 2 at study entry

  9. Life-expectancy of greater than 3 months

  10. Laboratory test results within these ranges at Screening and confirmed at enrollment prior to drug dosing on Cycle 1, Day 1:
* Absolute neutrophil count ≥ 1.5 x 10E9/L; if the bone marrow is extensively infiltrated ( ≥ 70% plasma cells) then ≥ 1.0 x 10E9/L
* Platelet count ≥ 75 x 10E9/L; if the bone marrow is extensively infiltrated ( ≥ 70% plasma cells) then ≥ 50 x 10E9/L patients must not have received platelet transfusion for at least 7 days prior to receiving screening platelet count. If patient have creatinine clearance of less than 60mL/min, patient's platelet count must be greater than 150 x 10E9/L.
* Hemoglobin ≥ 8.0 g/dL within 21 days prior to enrollment. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed; however, most recent RBC transfusion must have been at least 7 days prior to obtaining screening hemoglobin.
* Calculated or measured creatinine clearance (CrCl) of > 60 mL/minute (Study Part 1,2,3(2), and 4) or 30 to ≤ 60 mL/minute (Part 3(1)) as calculated by Cockcroft-Gault method (Appendix 3).
* Total bilirubin levels ≤ 2.0 mg/dL (normal levels)
* AST (SGOT) and ALT (SGPT) ≤ 2 x ULN
* Serum potassium 3.0 - 5.5 mEq/L

  11. Patients must be registered into the mandatory REVLIMID REMS™ program, and be willing and able to comply with the requirements of the REVLIMID REMS™ program

  12. FCBP† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting ruxolitinib and must either commit to continued abstinence from heterosexual intercourse or use acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, and at least 28 days before she starts taking ruxolitinib with or without lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

  † A FCBP (female of childbearing potential) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

  13. Able to take aspirin (acetylsalicylic acid, ASA) at 81 or 325 mg/daily as antiplatelet therapy if platelet count is above 30 x 10E9/L (subjects intolerant to ASA may use warfarin or low molecular weight heparin)

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria are not to be enrolled in the study:

  1. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
  2. Plasma cell leukemia (> 2.0 × 10E9/L circulating plasma cells by standard differential)
  3. Primary amyloidosis
  4. Non-hematologic malignancy within the past 5 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
  5. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

     * Myocardial infarction within 6 months prior to enrollment
     * New York Heart Association (NYHA) Class II or greater heart failure or uncontrolled angina
     * Clinically significant pericardial disease
     * Severe uncontrolled ventricular arrhythmias
     * Echocardiogram or MUGA evidence of LVEF below institutional normal within 28 days prior to enrollment
     * Electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
  6. Severe hypercalcemia, i.e., serum calcium ≥ 12 mg/dL (3.0 mmol/L) corrected for albumin
  7. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
  8. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
  9. Undergone major surgery within 28 days prior enrollment or has not recovered from side effects of such therapy (vertebroplasty or kyphoplasty is not considered to be a major surgery; however, the investigator is to discuss enrollment of a subject with a recent history of kyphoplasty with the medical monitor).
  10. Pregnant or breast feeding females (lactating females must agree not to breast feed while taking lenalidomide)
  11. Received the following prior therapy:

      * Chemotherapy within 3 weeks of study drugs
      * Corticosteroids (>20 mg/daily prednisone or equivalent) within 3 weeks of study drugs to ensure that steroid dose intensity at the beginning of the treatment is not altered by administration of steroids prior to the study. Consumption of steroids within 3 weeks of the treatment may interfere with efficacy and side effects due to differences of steroid intensity.
      * Immunotherapy or antibody therapy as well as thalidomide, arsenic trioxide, or bortezomib within 21 days before study drugs
      * Lenalidomide within 7 days before study drugs
      * Lenalidomide within 21 days before study drugs (Part 4 only)
      * Extensive radiation therapy within 28 days before study drugs. Receipt of localized radiation therapy does not preclude enrollment.
      * Use of any other experimental drug or therapy within 28 days of study drugs
      * Strong CYP3A4 inhibitors, strong CYP3A4 inducers and fluconazole doses >200 mg daily within 5 half-lives before study drugs. (For example, clarithromycin has half-life of 4 hours so washout period for clarithromycin is 20 hours.)
  12. Known hypersensitivity to compounds of similar chemical or biological composition to thalidomide and lenalidomide or steroids.
  13. Concurrent use of other anti-cancer agents or treatments
  14. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
  15. Known positivity for human immunodeficiency virus (HIV), hepatitis B or C, and /or active tuberculosis (TB) including subjects with latent TB or with the risk factor for activation of latent TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) of ruxolitinib in combination with steroids and lenalidomide [Tolerability]. | 30 months
  MTD will be determined by measuring incidence of the dose-limiting toxicities (DLTs) per dose level, of ruxolitinib in combination with steroids and lenalidomide for MM patients currently with progressive disease.
Incidence of Treatment-Emergent Adverse Events [Safety] | 54 months
  Safety will be measured by counting the occurrence of adverse events throughout the study, graded via Common Terminology Criteria for Adverse Events (CTCAE) v 4.03 criteria

SECONDARY OUTCOMES:
Overall response rate (ORR) as a measure of efficacy | 54 months
  Overall response rate (ORR) is defined as CR + VGPR + PR
Clinical benefit rate (CBR) as a measure of efficacy | 54 months
  Clinical benefit rate is defined as ORR + MR
Progression Free Survival (PFS) | 54 months
  Progression-free survival will be measured in months as the time from initiation of therapy to progressive disease or death from any cause, whichever occurs first
Assessment of the time to response as a measure of efficacy (TTR) | 54 months
  Time to response, defined as the time from the initiation of therapy to the first evidence of confirmed clinical benefit defined as > minimal response (MR, including patients who achieved a complete response (CR), very good partial response (VGPR), partial response (PR), or MR
Assessment of the duration of response as a measure of efficacy (DOR) | 54 months
  Duration of response, defined as the time (in months) from the first response to progressive disease
Assessment of the overall survival (OS) as a measure of efficacy | 54 months
  Overall survival, defined as the time (in months) from initiation of therapy to death from any cause or last follow-up visit
Assessment of the time to progression as a measure of efficacy (TTP) | 54 months
  Time to progression, defined as the time (in months) from the initiation of therapy to progressive disease.
Assessment of response in additional cohorts | 54 months
  Response to initial therapy (ruxolitinib and methylprednisolone alone) will be compared to the response to therapy with addition of lenalidomide (ruxolitinib, lenalidomide, methylprednisolone).
  Response to higher dose of ruxolitinib (20 mg BID) with steroids, the response will be compared to the initial response to therapy of patients treated with ruxolitinib (15 mg BID) alone with steroids as well as to the therapy with addition of lenalidomide (ruxolitinib, lenalidomide, methylprednisolone).

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (13):
- United States (13):
  - Global Oncology, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - California Cancer Associates for Research & Excellence (cCARE), Encinitas, California
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - Robert A. Moss, M.D., F.A.C.P., Inc., Fountain Valley, California
  - Pacific Cancer Care, Monterey, California
  - Sansum Clinic- Ridley-Tree Cancer Center, Santa Barbara, California
  - Wellness Oncology and Hematology, West Hills, California
  - James R. Berenson M.D. Inc., West Hollywood, California
  - Cancer Specialists, LLC, Jacksonville, Florida
  - Millennium Oncology Research Clinic, Pembroke Pines, Florida
  - Regional Cancer Care Associates (RCCA) MD, LLC, Bethesda, Maryland
  - Northwest Medical Specialists, PPLC, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berenson JR, Limon A, Rice S, Safaie T, Boccia R, Yang H, Moezi M, Lim S, Schwartz G, Eshaghian S, Brobeck M, Swift R, Eades BM, Bujarski S, Sebhat Y, Ray R, Kim S, Del Dosso A, Vescio R. A Phase I Trial Evaluating the Addition of Lenalidomide to Patients with Relapsed/Refractory Multiple Myeloma Progressing on Ruxolitinib and Methylprednisolone. Target Oncol. 2024 May;19(3):343-357. doi: 10.1007/s11523-024-01049-w. Epub 2024 Apr 20. PMID 38643346
- [Derived] Berenson JR, Martinez D, Safaie T, Boccia R, Yang H, Moezi M, Lim S, Schwartz G, Eshaghian S, Swift R, Eades BM, Bujarski S, Regidor B, Kim C, Kim S, Vescio R. Ruxolitinib and methylprednisolone for treatment of patients with relapsed/refractory multiple myeloma. Br J Haematol. 2023 Mar;200(6):722-730. doi: 10.1111/bjh.18593. Epub 2022 Dec 9. PMID 36482815
- [Derived] Berenson JR, Kim C, Bujarski S, To J, Spektor TM, Martinez D, Turner C, Ghermezi M, Eades BM, Swift RA, Schwartz G, Eshaghian S, Moss RA, Lim S, Vescio R. A phase 1 study of ruxolitinib, steroids and lenalidomide for relapsed/refractory multiple myeloma patients. Hematol Oncol. 2022 Dec;40(5):906-913. doi: 10.1002/hon.3066. Epub 2022 Aug 14. PMID 35946431
- [Derived] Berenson JR, To J, Spektor TM, Martinez D, Turner C, Sanchez A, Ghermezi M, Eades BM, Swift RA, Schwartz G, Eshaghian S, Stampleman L, Moss RA, Lim S, Vescio R. A Phase I Study of Ruxolitinib, Lenalidomide, and Steroids for Patients with Relapsed/Refractory Multiple Myeloma. Clin Cancer Res. 2020 May 15;26(10):2346-2353. doi: 10.1158/1078-0432.CCR-19-1899. Epub 2020 Jan 14. PMID 31937615